CLINICAL TRIAL: NCT02072148
Title: The Sinai Robotic Surgery Trial in HPV Positive Oropharyngeal Squamous Cell Carcinoma (SCCA)
Brief Title: The Sinai Robotic Surgery Trial in HPV Positive Oropharyngeal Squamous Cell Carcinoma (SCCA) (SIRS TRIAL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Raymond Chai, Associate Professor, Otolaryngology, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 13-1662
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Human Papilloma Virus; Oropharyngeal Squamous Cell Carcinoma
Keywords: Human Papilloma Virus; Oropharyngeal Squamous Cell Carcinoma; Transoral Robotic Surgery
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low Risk Group I (Experimental): Group I:
  * Complete resection (margins: tonsil >1mm, tongue >3mm, pT1-2, pN0-2B),
  * No LVI, no PNI, <3 positive nodes.
  * No ECS, No matted or Level >III,
  Interventions: Procedure: PET/CT
- Intermediate Risk Group II (Experimental): Group II
  * Complete resection (margins: tonsil <1mm, tongue <1mm, pT1-2, pN0-2B),
  * +LVI, +PNI, <3 positive nodes. ≤1mm ECS.
  Interventions: Procedure: PET/CT; Radiation: Radiotherapy
- High Risk Group IIIA (Experimental): * 3+ nodes, no ECS > 1mm
  * Contralateral or supraclavicular nodes
  Interventions: Procedure: PET/CT; Radiation: Concurrent Chemoradiation
- High Risk Group IIIB (Experimental): * Incomplete surgical resection with + surgical margins
  * ≥ 1 mm ECS
  * Matted nodes
  Interventions: Procedure: PET/CT; Radiation: Concurrent Chemoradiation

INTERVENTIONS:
Procedure: PET/CT — PET scan or CT scan q 4 months for 5 years
Radiation: Radiotherapy — Postoperative XRT 5000 cGy
  Other Names: RT; XRT
  Arms: Intermediate Risk Group II
Radiation: Concurrent Chemoradiation — CCRT with cisplatin 40mg/m2/week IV over approximately 30 minutes, mixed in 250ml normal saline Weekly on Monday or Tuesday any time, or Wednesday prior to radiation
  Postoperative XRT 5000 cGy
  Other Names: CCRT; Cisplatin
  Arms: High Risk Group IIIA
Radiation: Concurrent Chemoradiation — CCRT with cisplatin 40mg/m2/week IV over approximately 30 minutes, mixed in 250ml normal saline Weekly on Monday or Tuesday any time, or Wednesday prior to radiation
  Postoperative XRT 5600 cGy
  Other Names: CCRT; Cisplatin
  Arms: High Risk Group IIIB

SUMMARY:
In general, patients with Human Papilloma Virus Positive Oropharyngeal Squamous Cell Carcinoma (HPVOPC) are curable, young and will live for prolonged periods. They are at high risk for long-term toxicity and mortality from therapy. While the long-term consequences of chemotherapy and surgery for head and neck cancer are relatively constrained, high-dose radiotherapy (RT) and chemoradiotherapy (CRT) substantially impact on local tissues and organ function and result in a significant rate of late mortality and morbidity in patients. Studies are now being designed to reduce the impact of RT and CRT for patients.

Patients with intermediate stage HPV positive oropharyngeal cancer will be screened for poor prognostic features and undergo robotic surgery. Patients in whom pathology demonstrates good prognosis features will then be followed without postoperative radiotherapy. Patients with subsequent recurrence will be treated with either surgery and postoperative radiotherapy or postoperative chemoradiotherapy alone. Patients with poor prognostic features (ECS, LVI, PNI) will receive reduced dose radiotherapy or chemoradiotherapy based on pathology. It is expected that over 50% of patients treated with surgery will have had a curative treatment and will avoid radiation therapy entirely and long-term survival will not be changed by withholding radiation therapy to good prognosis patients after surgery. There are exploratory biomarkers of risk of recurrence that will be collected and studied.

There are currently few trials examining the role of de-escalation using surgery alone in intermediate and early T-stage HPV related disease. New surgical techniques have broadened the range of patients capable of achieving a complete resection and the functional outcomes in such patients are outstanding. Furthermore, the sensitivity of HPVOPC to chemotherapy and radiotherapy raise the possibility that delayed or salvage treatment in early stage patients would be highly effective, would result in similar survival outcomes and radiotherapy could be applied to a much smaller population then current standards call for. Looked at from a different perspective, the need for post-operative radiotherapy in this younger, HPV+ and more functional population has not been validated in clinical trials to date.

ELIGIBILITY:
Inclusion Criteria:

* Patients may be screened and consented if they display clinical features that are consistent with p16 positivity, they are p16+ but and not yet tested for p16 by IHC and for HPV by PCR and if they meet the other eligibility criteria. They will enter the experimental post-surgical portion of the study if they have surgery performed at MSSM and surgical specimens or biopsies proven to be both p16+ on IHC testing and HPV+ on PCR testing
* Participants must have histologically or cytologically confirmed and identified resectable primary squamous cell carcinoma of the oropharynx that is HPV 16 positive or positive for any high risk HPV subtype (i.e., 18, 33, 35, etc.) as determined by PCR at the central laboratory. Patients must have p16+ status as determined by IHC performed or reviewed at the central laboratory prior to consent. Both p16 and HPV status must be determined prior to post-surgical adjuvant treatment assignment. Tissue from the primary site must be available for biomarker studies after surgery.
* Stage 1, 2, 3 or early and intermediate stage IVa (T1N0-2B, T2N0-2B) (Level 2, non-matted) disease without evidence distant metastases or extracapsular extension. Primary site must be lateralized for a functional dissection.
* Age > 18 years.
* No previous surgery, radiation therapy or chemotherapy for SCCHN (other than biopsy or tonsillectomy) is allowed at time of study entry.
* ECOG performance status of 0 or 1.
* No active alcohol addiction (as assessed by medical caregiver).
* No active tobacco use (>10 years tobacco free interval, <20pk/yr. history)
* Ability to understand and the willingness to sign a written informed consent document.
* Participants must have adequate bone marrow, hepatic and renal functions as defined below:

  1. Hematology:

     * Neutrophil count > 1.5 x 109/l.
     * Platelet count > 100 x 109/l.
     * Hemoglobin > 10 g/dl (may achieve by transfusion).
  2. Renal function: > 60 ml/min (actual or calculated by the Cockcroft-Gault method) as follows:

     * CrCl (mL/min) = (140-age) (weight kg)
     * 72 x serum creatinine (mg/dL)
     * N.B. For females, use 85% of calculated CrCl value.
     * Or a Creatinine < the upper limits of normal

Exclusion Criteria:

* Patients < age 18.
* Pregnant or breast feeding women.
* Previous or current malignancies at other sites, with the exception of adequately treated in situ carcinoma of the cervix, basal or squamous cell carcinoma of the skin, thyroid cancer, or other cancer curatively treated by surgery and with no current evidence of disease for at least 5 years.
* Other serious illnesses or medical conditions including but not limited to:

  1. Unstable cardiac disease despite treatment, myocardial infarction with months prior to study entry.
  2. History of significant neurologic or psychiatric disorders including dementia or seizures
  3. Active clinically significant uncontrolled infection
  4. Active peptic ulcer disease defined as unhealed or clinically active
  5. Active drug addiction including alcohol, cocaine or intravenous drug use defined as occurring within the 6 months preceding diagnosis
  6. Chronic Obstructive Pulmonary Disease, defined as being associated with a hospitalization for pneumonia or respiratory decompensation within 12 months of diagnosis. This does not include obstruction from tumor
  7. Autoimmune disease requiring therapy, prior organ transplant, or known HIV infection
  8. Interstitial lung disease
  9. Hepatitis C by history
  10. Concurrent treatment with any other anticancer therapy.
  11. Participation in an investigational therapeutic drug trial within 30 days of study entry.
* Advanced Stage III,IV (N2C, N3) or surgically unresectable disease or disease that cannot be fully resected, obvious radiologic ECS, supraclavicular or matted metastatic disease, >3 cervical nodes. (These patients will be placed on the Quarterback trial due to advanced state of disease and poor prognostic features)
* HPV negative OPSCC as determined by determined by PCR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2014-03; Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Posner, MD, Study Director — Icahn School of Medicine at Mount Sinai; Raymond Chai, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Mount Sinai Beth Israel, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 112 participants enrolled prior to transoral surgery. 63 were evaluable and assigned to arm based on risk.
Groups:
- Low Risk Group I: Group I:
  * Complete resection (margins: tonsil >1mm, tongue >3mm, pT1-2, pN0-2B),
  * No LVI, no PNI, <3 positive nodes.
  * No ECS, No matted or Level >III,
  Observation
- Intermediate Risk Group II: Group II
  * Complete resection (margins: tonsil <1mm, tongue <1mm, pT1-2, pN0-2B),
  * +LVI, +PNI, <3 positive nodes. ≤1mm ECS.
  Radiotherapy: Postoperative XRT 50 Gy
- High Risk Group III: IIIA
  * 3+ nodes, no ECS > 1mm
  * Contralateral or supraclavicular nodes
  IIIB:
  * Incomplete surgical resection with + surgical margins
  * ≥ 1 mm ECS
  * Matted nodes
  Concurrent Chemoradiation: CCRT with cisplatin 40mg/m2/week IV over approximately 30 minutes, mixed in 250ml normal saline Weekly on Monday or Tuesday any time, or Wednesday prior to radiation
  Postoperative XRT 56 Gy
Period: Overall Study
Arm/Group | Low Risk Group I | Intermediate Risk Group II | High Risk Group III
Started | 54 | 29 | 29
Completed | 31 | 16 | 16
Not Completed | 23 | 13 | 13
Not completed — withdrew prior to surgery | 23 | 0 | 0
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Risk Group I | Intermediate Risk Group II | High Risk Group III | Total
Number analyzed (Participants) | 54 | 29 | 29 | 112
Age, Continuous [Mean (Full Range); unit: years] | 62 [42 to 84] | 68 [54 to 79] | 70 [56 to 81] | 66 [42 to 84]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 50 | 20 | 26 | 96
  Gender: Female | 4 | 9 | 3 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Disease Specific Survival (DSS)
Description: Number of participants with HPV related oropharynx cancer treated with a de-intensified adjuvant protocol with status of disease specific survival. DSS was calculated by measuring the time from trial entry to cancer-related death.
Time Frame: 5 years
Measure: Number; unit: participants
Groups:
- Intermediate Risk Group II: Group II
  * Complete resection (margins: tonsil <1mm, tongue <1mm, pT1-2, pN0-2B),
  * +LVI, +PNI, <3 positive nodes. ≤1mm ECS.
  Radiotherapy: Postoperative XRT 50 Gy in 25 fractions
- High Risk Group III: IIIA
  * 3+ nodes, no ECS > 1mm
  * Contralateral or supraclavicular nodes
  IIIB:
  * Incomplete surgical resection with + surgical margins
  * ≥ 1 mm ECS
  * Matted nodes
  Concurrent Chemoradiation: CCRT with cisplatin 40mg/m2/week IV over approximately 30 minutes, mixed in 250ml normal saline Weekly on Monday or Tuesday any time, or Wednesday prior to radiation
  Postoperative XRT 56 Gy in 28 fractions
Arm/Group | Low Risk Group I | Intermediate Risk Group II | High Risk Group III
Number analyzed (Participants) | 31 | 16 | 16
participants | 29 | 15 | 15

2. Primary Outcome: Number of Participants With Progression-Free Survival (PFS)
Description: Number of participants with HPV related oropharynx cancer treated with a de-intensified adjuvant protocol with status of progression-free survival. PFS calculated the time to biopsy confirmed recurrence or death from any cause.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk Group I | Intermediate Risk Group II | High Risk Group III
Number analyzed (Participants) | 31 | 16 | 16
Participants | 29 | 15 | 15

3. Primary Outcome: Number of Participants With Locoregional Failures (LRFs)
Description: the rate of local regional control (LRC) in patients with early and intermediate stage HPV related oropharynx cancer treated with surgery alone as assessed by number of participants with locoregional failures.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk Group I | Intermediate Risk Group II | High Risk Group III
Number analyzed (Participants) | 31 | 16 | 16
Participants | 29 | 15 | 15

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) in patients with early and intermediate stage HPV related oropharynx cancer treated with surgery alone. OS from the time of entry to death with any cause.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk Group I | Intermediate Risk Group II | High Risk Group III
Number analyzed (Participants) | 31 | 16 | 16
Participants | 31 | 16 | 15

5. Secondary Outcome: Number of Serious Adverse Events
Description: Number of serious adverse events
Time Frame: 5 years
Measure: Number; unit: events
Arm/Group | Low Risk Group I | Intermediate Risk Group II | High Risk Group III
Number analyzed (Participants) | 31 | 16 | 16
events | 1 | 0 | 2

6. Secondary Outcome: Global Quality of Life Scores
Description: Global Quality of Life Scores total score from 0-100, with higher score indicating better health outcomes.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: score on a scale (MDADI score)
Arm/Group | Low Risk Group I | Intermediate Risk Group II | High Risk Group III
Number analyzed (Participants) | 31 | 16 | 16
score on a scale (MDADI score)
  baseline, prior to surgery | 89 (5) | 89 (4) | 89 (12)
  3 months | 89 (6) | 76 (6) | 63 (10)
  6 months | 89 (4) | 85 (4) | 71 (13)
  1 year | 89 (4) | 85 (6) | 78 (9)
  2 years | 89 (3) | 85 (6) | 88 (9)

ADVERSE EVENTS:
Time Frame: 5 years
Description: Definitions do not differ from clinical.trials.gov definitions.
Arm/Group | Low Risk Group I | Intermediate Risk Group II | High Risk Group III
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/16 | 1/16
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/16 | 2/16
Other Adverse Events (participants affected / at risk) | 15/31 | 16/16 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Risk Group I (N=31) | Intermediate Risk Group II (N=16) | High Risk Group III (N=16)
Bleeding (Blood and lymphatic system disorders) | 1 | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Risk Group I (N=31) | Intermediate Risk Group II (N=16) | High Risk Group III (N=16)
dysphagia (General disorders) | 10 | 0 | 16
severe pain (General disorders) | 8 | 10 | 16
anxiety (Psychiatric disorders) | 3 | 0 | 0
xerostomia (General disorders) | 3 | 10 | 0
postoperative bleed (Surgical and medical procedures) | 1 | 0 | 1 — requiring operative management
velopharyngeal insufficiency (Surgical and medical procedures) | 1 | 0 | 0
altered taste/dysgeusia (General disorders) | 0 | 15 | 0
numbness of the neck (Surgical and medical procedures) | 0 | 3 | 0
lack of appetite (General disorders) | 0 | 3 | 0
dysarthria (General disorders) | 0 | 0 | 8
mucositis (General disorders) | 0 | 0 | 15
>20-lb weight loss (Metabolism and nutrition disorders) | 0 | 0 | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
hematoma (Surgical and medical procedures) | 0 | 0 | 1 — requiring operative management
neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 3
thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3
dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
tinnitus (Ear and labyrinth disorders) | 0 | 0 | 2
creatinine elevation (Renal and urinary disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Small sample size within each group limiting the generalizability of the reported results. The mean length of follow-up (43.8 months) is shorter than the standard 5-year reporting criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT02072148/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT02072148/ICF_001.pdf